CLINICAL TRIAL: NCT05800080
Title: An Exploratory Study of Immunotherapy Combined With Anlotinib Hydrochloride Capsules and Chemotherapy in Perioperative Treatment of Locally Advanced Novel Coronavirus Infected Gastric Cancer
Brief Title: An Exploratory Study of Immunotherapy Combined With Anlotinib and Chemotherapy in Perioperative Treatment of LAGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-W-0031
Record Dates: First submitted 2023-02-16; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: one group receives peri operative treatment of Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy, and the other group receives peri operative treatment of Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy Penpulimab (single immunity, fixed dose 200mg) orCadonilimab (double immunity, fixed dose 500mg), which will be administered on the first day of each cycle and repeated every three weeks; Anlotinib Hydrochloride Capsules: 12mg, administered on the 1-14th day of each cycle
  Other Names:
  Teggio Oxaliplatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single immunotherapy group； (Experimental): one group receives peri operative treatment of Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy；
  Interventions: Drug: Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy;Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy
- Double immune treatment group (Experimental): one group receives peri operative treatment of Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy
  Interventions: Drug: Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy;Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy

INTERVENTIONS:
Drug: Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy;Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy — one group receives peri operative treatment of Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy, and the other group receives peri operative treatment of Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy.After receiving corresponding neoadjuvant treatment for 3 cycles according to the established treatment plan, surgical treatment shall be carried out within 3-6 weeks after drug withdrawal
  Other Names: Teggio; Oxaliplatin

SUMMARY:
* 1. Main objective: to evaluate the pathological complete response (pCR) of gastric cancer after local advanced COVID-19 infection by two kinds of immunotherapy combined with Anlotinib Hydrochloride Capsules and neoadjuvant chemotherapy.
* 2. Secondary objective: to evaluate the major pathological response (MPR), disease-free survival (DFS), objective response rate (ORR), R0 resection rate (R0 resection rate) and safety of two kinds of immunotherapy combined with Anlotinib Hydrochloride Capsules and neoadjuvant chemotherapy for gastric cancer after local advanced COVID-19 infection。

DETAILED DESCRIPTION:
This is a prospective multicenter exploratory study to evaluate the efficacy and safety of two kinds of immunotherapy combined with Anlotinib Hydrochloride Capsules and chemotherapy for resectable or potentially resectable T3~4N+M0 locally advanced gastric cancer after COVID-19 infection This study was led by Professor Hongliu, Department of Gastroenterology, Xijing Hospital. 114 patients with resectable or potentially resectable T3~4N+M0 locally advanced gastric cancer were planned to be randomly divided into two groups: one group received peri-operative treatment with Penpulimab combined with Anlotinib Hydrochloride Capsules and chemotherapy, and the other group received peri-operative treatment with Cadonilimab combined with Anlotinib Hydrochloride Capsules and chemotherapy. Each subject will receive three cycles of neoadjuvant study treatment: Pianzumab (single immunity, fixed dose 200mg) or Cadonilimab (double immunity, fixed dose 500mg), which will be administered on the first day of each cycle and repeated every three weeks; Anlotinib Hydrochloride Capsules: 12mg, administered on the 1-14th day of each cycle, once a day, about half an hour before breakfast (the time of daily administration should be the same as much as possible), delivered with warm water, repeated once every 3 weeks; Tegafur: It needs to be administered according to the patient's body surface area< 40 mg/time at 1.25 m2; ≥ 50 mg/time when 1.25m2 and<1.5 m2; ≥ 60 mg/time at 1.5 m2; Take orally, twice a day, after breakfast and dinner, for 14 consecutive days, and rest for 7 days, which is a treatment cycle; Repeat once every 3 weeks; Oxaliplatin: 130 mg/m2, administered on the first day of each cycle, repeated every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 70 years old, male or female;
* ECOG score 0-1 points;
* Patients with locally advanced gastric cancer confirmed by pathology (histology or cytology) (according to WHO classification in 2015);
* Nucleic acid test or antigen test to identify patients with COVID-19 infection
* According to the TNM stage of clinical tumor in the 8th edition, T3~4N+M0 gastric cancer patients confirmed as resectable or potentially resectable by endoscopic ultrasound and enhanced CT;
* It has measurable lesions (according to RECIST 1.1 standard, the long diameter of CT scan of tumor lesions is ≥ 10mm, and the short diameter of CT scan of lymph node lesions is ≥ 15mm;);
* Those who were diagnosed as gastric cancer for the first time before enrollment and did not undergo radiotherapy, chemotherapy, surgery and targeted treatment;
* The function of main organs is normal, that is, they meet the following standards:
* The blood routine examination must meet the following requirements (no blood transfusion, no hemopoietic factor and no drug correction within 14 days):
* ANC ≥ 1.5 × 109/L；
* PLT ≥ 100 × 109/L；
* HB ≥ 90 g/L；
* Biochemical examination shall meet the following standards:
* TBIL≤1.5 × ULN；
* ALT、AST≤ 2.5 × ULN
* Serum creatinine sCr ≤ 1.5 × ULN, endogenous creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula);
* Coagulation function must meet: INR ≤ 1.5 × ULN and APTT ≤ 1.5 × ULN；
* Female subjects of childbearing age must carry out a serum pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved effective contraceptive measure (such as intrauterine device, contraceptive or condom) during the study period and within 3 months after the last administration of the study medication; For male subjects whose partners are women of childbearing age, they should undergo surgical sterilization or agree to use effective methods of contraception during the study and within 3 months after the last study administration;
* Subjects voluntarily joined the study and signed the informed consent form, with good compliance and cooperation in follow-up;

Exclusion criteria:

* Patients with distant metastasis;
* Subjects who have previously received anti-PD-1 (L1) or CTLA4 monoclonal antibodies;
* Medical history and complications
* Other malignant tumors in the past 3 years;
* Have any history of active autoimmune diseases or autoimmune diseases (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy); Patients with vitiligo or childhood asthma have been completely relieved and can be included without any intervention after adulthood; Patients who need bronchodilator for medical intervention cannot be included;
* Immunosuppressive drugs were used within 14 days before the first use of the study drug, excluding nasal spray and inhaled corticosteroids or systemic steroid hormones with physiological dose (i.e. no more than 10 mg/day prednisone or its equivalent);
* Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite the best drug treatment);
* Newly diagnosed angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; Arrhythmias (including QTcF: male ≥ 450 ms, female ≥ 470 ms) require long-term use of antiarrhythmic drugs and cardiac insufficiency of New York Heart Association grade ≥ II; Or uncontrolled heart failure;
* There is evidence that there is pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia and serious damage to lung function in the past or at present;
* Severe infection (such as the need for intravenous drip of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or fever of unknown cause occurred during screening/before the first administration>38.5 ° C;
* There is clinically significant hemoptysis (more than 50 mL of hemoptysis per day) within the first three months of the study, or there is clinically obvious bleeding symptom or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood++or above the baseline, or suffering from vasculitis).
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Inoculate live attenuated vaccine within 4 weeks before the first administration or during the study period;
* Physical examination and laboratory examination findings
* People with congenital or acquired immune deficiency, such as people infected with human immunodeficiency virus (HIV), active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the detection limit of the analytical method) or combined with hepatitis B and hepatitis C infection;
* Pregnant or lactating women; Those with fertility who are unwilling or unable to take effective contraceptive measures;
* Known to have a positive history of human immunodeficiency virus (HIV) test or known to have acquired immunodeficiency syndrome (AIDS);
* Allergic reactions, allergic reactions and adverse drug reactions
* Severe allergic reaction to other monoclonal antibodies;
* Allergy or intolerance to infusion;
* Have a history of severe allergy to arotinib or its preventive drugs;
* Subjects who are participating in other clinical studies or whose first medication is less than 4 weeks from the end of the previous clinical study (the last medication), or who have 5 half-lives of the study drug;
* Subjects are known to have a history of abuse of psychotropic substances, alcohol abuse or drug abuse;
* The researcher believes that there are any conditions that may damage the subject or cause the subject to fail to meet or perform the research requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response; | 12months
  Defined as tumor tissue specimens resected surgically after neoadjuvant therapy with no residual tumor cells.

SECONDARY OUTCOMES:
major pathologic response, MPR | 12months
  Defined as tumor specimens resected after neoadjuvant therapy with residual tumor cells ≤10%

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, Study Chair — Air Force Military Medical University, China
Locations (1):
- The First Affiliated Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No